CLINICAL TRIAL: NCT04633850
Title: Implementation of Adjuvants in Intercostal Nerve Blockades for Thoracoscopic Surgery in Pulmonary Cancer Patients: A Before and After Study
Brief Title: Implementation of Adjuvants in Intercostal Nerve Blockades for Thoracoscopic Surgery in Pulmonary Cancer Patients
Status: Completed | Type: Observational
Sponsor: Jannie Bisgaard Stæhr (Other)
Responsible Party: Sponsor-Investigator, Jannie Bisgaard Stæhr, MD PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: Smerter efter VATS
Record Dates: First submitted 2020-11-03; First posted 2020-11-18 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain; Lung Cancer; Video Assisted Thoracoscopic Surgery; Thoracoscopic Surgery; Nerve Block; Local Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Lung Neoplasms | interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before implementation: Perineural bupivacaine without adjuvants.
  Interventions: Drug: Bupivacain
- After implementation: Perineural bupivacaine with intravenous dexamethasone.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Intravenous dexamethasone 8 mg. Given once at the end of surgery.
  Groups: After implementation
Drug: Bupivacain — Bupivacaine dose according to weight. <60 kg: Total dose 100mg 60-90kg: Total dose 150mg >90kg: Total dose 200mg
  Given once at the end of surgery.
  Groups: Before implementation

SUMMARY:
To investigate the effect of intercostal blockade with and without adjuvants.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive routine procedure. It's less invasive than thoracotomy but postoperative pain is still a problem.

At Aalborg University Hospital, intercostal blockades with bupivacaine is used as standard pain treatment for patients undergoing VATS. Adding adjuvants to the blockades may prolong the effect.

The aim of this study is to investigate if intercostal nerve blockade with adjuvants (intravenous (IV) dexamethasone) will result in better pain management.

The primary plan was to evaluate the effect of adding IV dexamethasone and perineural adrenaline, but due to adverse effects, adrenaline was first reduced and later removed from the intervention (amendment protocol N-20200040 approved by the Ethics Committee of Northern Jutland on February 2nd 2021).

ELIGIBILITY:
Inclusion Criteria:

° Consecutive adult patients over 18 years of age scheduled to undergo VATS because of verified/suspected lung cancer.

Exclusion Criteria:

* Inability to understand verbal and written information.
* Preexisting chronic pain condition.
* Preoperative daily treatment with pain medication (Non-opioids, opioids, gabapentin/pregabalin).
* Previous thoracic surgery.
* Previous chemotherapy due to thoracic malignancy and / or radiation therapy. to the thorax.
* Pregnant women.
* Autoimmune neuromuscular diseases (sclerosis, peripheral neuromuscular disorders). General muscle weakness or atrophy.
* Hypersensitivity, allergy or intolerance to dexamethasone, bupivacaine or adrenaline.
* Preoperative epidural anaesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lung cancer patients scheduled to undergo VATS at Aalborg University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Total equipotent dose of opioids | 24 hours
  Sum of equipotent opioid doses during the first 24 hours after surgery

SECONDARY OUTCOMES:
Time to first administration of opioids after surgery | 48 hours
  In hours and minuts
Numerical rating scale score | 24 hours
  Pain score reported by the patient after surgery from 0 (no pain) to 10 (worst imaginable pain) in whole numbers.
Time for full mobilization | Through study completion, an average of 1 week
  The total time for full mobilization (walk with support)
Total dose of non-opioid analgesics | 24 hours
  Sum of non-opioid doses during the first 24 hours after surgery
The need for pain medication at discharge | At discharge from hospital, an average of 1 week
  The need for pain medication at discharge (all forms, type, dose)
Postoperative complication (Empyema) | At discharge from hospital, an average of 1 week
  Empyema (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)
Postoperative complication (Air leakage) | At discharge from hospital, an average of 1 week
  Air leakage (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)
Postoperative complication (Reoperation) | At discharge from hospital, an average of 1 week
  Reoperation (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)
Postoperative complication (Pneumonia) | At discharge from hospital, an average of 1 week
  Pneumonia (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)
Postoperative complication (Drainage of pleural effusion) | At discharge from hospital, an average of 1 week
  Pleural effusion (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)
Postoperative complication (Oyxgen therapy) | At discharge from hospital, an average of 1 week
  The need for supplemental oxygen therapy and need for mechanical ventilation (yes/no) as complication to the surgery described in the patients journal at discharge (epicrisis)

CONTACTS AND LOCATIONS:
Overall Officials: Jannie Bisgaard Stæhr, PhD, MD, Principal Investigator — Department of Anaesthesia
Locations (1):
- Aalborg University Hospital, Aalborg, Region of Northern Jutland, Denmark

REFERENCES:
- [Derived] Lobel J, Danielsen AV, Sperling PK, Bisgaard J. Intravenous dexamethasone in pain treatment after video-assisted thoracoscopic surgery. Dan Med J. 2024 Feb 12;71(3):A05230317. doi: 10.61409/A05230317. PMID 38445317